CLINICAL TRIAL: NCT00830557
Title: Biospecimen Resource for Pancreas Research, a Data & Tissue Bank (Also Known as a Bio-repository, Bio-bank, Data & Tissue Database, Data & Tissue Registry, Etc.) to Help Advance Research in Pancreas Disease
Brief Title: Collecting Medical Information and Tissue Samples From Patients With Pancreatic Cancer or Other Pancreatic Disorders
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shounak Majumder, Principal Investigator, Mayo Clinic
Other Study IDs: 354-06; P50CA102701-08 (NIH); CDR0000613100 (Other: NCI)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Islet Cell Tumor; Pancreatic Cancer; Pancreatic Disease; Acute Pancreatitis; Chronic Pancreatitis; Hereditary Pancreatitis; Pancreatic Neuroendocrine Carcinoma
Keywords: recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent islet cell carcinoma; pancreatic alpha cell carcinoma; pancreatic beta islet cell carcinoma; pancreatic delta cell carcinoma; pancreatic G-cell carcinoma
MeSH Terms: conditions — Adenoma, Islet Cell; Pancreatic Neoplasms; Pancreatic Diseases; Pancreatitis; Pancreatitis, Chronic; Hereditary pancreatitis; Somatostatinoma; Carcinoma, Islet Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Two 10mL plasma tubes, two 10mL serum tubes and one 10mL heparin tube collected. DNA extracted from lymphocytes. Possible saliva collection for DNA extraction. Waste tissue from prior surgery may be collected. Stool samples may be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: Patients undergo blood, saliva, and previously obtained leftover tissue sample collection on study. Patients also complete questionnaires and have their medical records reviewed on study.
  Interventions: Other: medical chart review; Other: survey administration; Other: biospecimen collection

INTERVENTIONS:
Other: medical chart review — baseline, 12 month and 36 months
Other: survey administration — baseline, 6 month, 12 month
Other: biospecimen collection — baseline

SUMMARY:
RATIONALE: Gathering medical information and collecting and storing samples of blood and tissue to test in the laboratory may help doctors develop better ways to screen people at risk for pancreatic cancer or other pancreatic disorders in the future.

PURPOSE: This clinical trial is collecting medical information and tissue samples from patients with pancreatic cancer or other pancreatic disorders.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To maintain a resource (bank) of biospecimens and data collected from individuals being seen clinically for pancreas conditions to facilitate the discovery and development of (but not limited to) biomarkers of risk (including genomic and proteomic) and early detection as well as novel targeted therapies for pancreatic diseases with a focus on pancreatic cancer.

OUTLINE: This is an observational study.

Patients undergo blood, saliva, and previously obtained leftover tissue sample collection on study. Patients also complete questionnaires and have their medical records reviewed on study.

ELIGIBILITY:
* Known or suspected pancreas disease including:

  * pancreas adenocarcinoma
  * islet cell cancer
  * pancreatic cysts
  * pancreatitis (hereditary, acute, or chronic)
* Next of kin of deceased participant who did not complete participation before passing away

Exclusion Criteria:

* Under the age of 18
* Unable to provide informed consent
* Prison inmates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected pancreas disease including pancreas adenocarcinoma, islet cell cancer, pancreatic cysts, pancreatitis (hereditary, acute, or chronic) or the next of kin of deceased participants.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2000-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Collection of clinical data, health and family histories by survey | baseline enrollment, 6 months, 12 months
Collection of blood and/or tissue, fecal and oral specimens | baseline
Collection of information regarding food preparation and intake by survey | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shounak Majumder, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials